CLINICAL TRIAL: NCT00862654
Title: Efficacy and Safety of Clobetasol Propionate Shampoo 0.05% Used in Association With an Antifungal Shampoo in the Treatment of Moderate to Severe Scalp Seborrheic Dermatitis
Brief Title: Clobetasol Propionate 0.05% Shampoo in Association With Antifungal Shampoo in Scalp Seborrheic Dermatitis
Acronym: Escape
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.29079
Record Dates: First submitted 2009-03-15; First posted 2009-03-17 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2011-08

CONDITIONS: Scalp Seborrheic Dermatitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- C propionate 4/week + Ketoconasole 2/week (Experimental): Clobetasol propionate shampoo 0.05% (4/week) + Ketoconazole shampoo 2% (2/week)
  Interventions: Drug: clobetasol propionate shampoo (4/week) - ketoconazole shampoo (2/week)
- C propionate 2/week + Ketoconasole 2/week (Experimental): Clobetasol propionate shampoo 0.05% (2/week) + Ketoconazole shampoo 2% (2/week)
  Interventions: Drug: clobetasol propionate shampoo (2/week) - ketoconazole shampoo (2/week)
- C propionate 2/week (Experimental): Clobetasol propionate shampoo 0.05% (2/week)
  Interventions: Drug: clobetasol propionate shampoo (2/week)
- Ketoconazole 2/week (Active Comparator): Ketoconazole shampoo 2% (2/week)
  Interventions: Drug: ketoconazole shampoo (2/week)

INTERVENTIONS:
Drug: clobetasol propionate shampoo (4/week) - ketoconazole shampoo (2/week) — Association: clobetasol propionate shampoo & ketoconazole shampoo
  Arms: C propionate 4/week + Ketoconasole 2/week
Drug: clobetasol propionate shampoo (2/week) - ketoconazole shampoo (2/week) — Association: clobetasol propionate shampoo & ketoconazole shampoo
  Arms: C propionate 2/week + Ketoconasole 2/week
Drug: clobetasol propionate shampoo (2/week) — Monotherapy with clobetasol propionate shampoo
  Arms: C propionate 2/week
Drug: ketoconazole shampoo (2/week) — Monotherpay ketoconazole shampoo (2/week)
  Arms: Ketoconazole 2/week

SUMMARY:
The objective is to assess different treatment regimens with Clobetasol propionate shampoo 0.05% in the treatment of scalp Seborrheic Dermatitis.

DETAILED DESCRIPTION:
The objective is to assess different treatment regimens with Clobetasol propionate shampoo 0.05% in association with an antifungal shampoo (Ketoconazole 2%) in the treatment of moderate to severe scalp Seborrheic Dermatitis compared to the antifungal shampoo alone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate to severe scalp Seborrheic Dermatitis

Exclusion Criteria:

* Subjects suffering from psoriasis,
* Subjects with a known allergy to one of the components of the test products,
* Female subjects who are pregnant, nursing or planning a pregnancy during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Ortonne, MD, Principal Investigator — Nice Hospital (France)
Locations (18):
- Belgium (6):
  - Galderma Investigational Center, Bruges
  - Galderma Investigational Center, Brussels
  - Galderma Investigational Center, Geel
  - Galderma Investigational Center, Ghent
  - Galderma Investigational Center, Liège
  - Galderma Investigational Center, Mons
- Galderma Investigational Center, Paris, France
- Germany (6):
  - Galderma Investigational Center, Berlin
  - Galderma Investigational Center, Bonn
  - Galderma Investigational Center, Hamburg
  - Galderma Investigational Center, Lübeck
  - Galderma Investigational Center, Mahlow
  - Galderma Investigational Center, Wuppertal
- Mexico (4):
  - Galderma Investigational Center, Guadalajara
  - Galderma Investigational Center, México
  - Galderma Investigational Center, Naucalpan
  - Galderma Investigational Center, Zapopan, Jalisco
- Galderma Investigational Center, Seoul, South Korea

REFERENCES:
- [Derived] Ortonne JP, Nikkels AF, Reich K, Ponce Olivera RM, Lee JH, Kerrouche N, Sidou F, Faergemann J. Efficacious and safe management of moderate to severe scalp seborrhoeic dermatitis using clobetasol propionate shampoo 0.05% combined with ketoconazole shampoo 2%: a randomized, controlled study. Br J Dermatol. 2011 Jul;165(1):171-6. doi: 10.1111/j.1365-2133.2011.10269.x. PMID 21707573
- See also: Sponsor general information — http://www.galderma.com

RESULTS

PARTICIPANT FLOW:
Groups:
- C Propionate 4/Week + Ketoconazole 2/Week: Clobetasol propionate shampoo 0.05% (4/week) + Ketoconazole shampoo 2% (2/week)
- C Propionate 2/Week + Ketoconazole 2/Week: Clobetasol propionate shampoo 0.05% (2/week) + Ketoconazole shampoo 2% (2/week)
- Ketakonazol 2/Week: Ketoconazole shampoo 2% (2/week)
Period: Overall Study
Arm/Group | C Propionate 4/Week + Ketoconazole 2/Week | C Propionate 2/Week + Ketoconazole 2/Week | C Propionate 2/Week | Ketakonazol 2/Week
Started | 82 | 82 | 82 | 80
Completed | 76 | 74 | 76 | 74
Not Completed | 6 | 8 | 6 | 6
Not completed — Lack of Efficacy | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1 | 3
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Pregnancy | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 2 | 3
Not completed — Subject mistake | 0 | 1 | 0 | 0
Not completed — Familly constraint | 0 | 1 | 0 | 0
Not completed — Never used study drugs | 1 | 0 | 0 | 0
Not completed — Included after end of inclusions | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | C Propionate 4/Week + Ketoconazole 2/Week | C Propionate 2/Week + Ketoconazole 2/Week | C Propionate 2/Week | Ketakonazol 2/Week | Total
Number analyzed (Participants) | 82 | 82 | 82 | 80 | 326
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3 | 1 | 7
  Between 18 and 65 years | 65 | 69 | 71 | 66 | 271
  >=65 years | 15 | 12 | 8 | 13 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (16.0) | 43.8 (17.2) | 44.9 (15.3) | 44.7 (15.5) | 45.1 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 39 | 38 | 36 | 149
  Male | 46 | 43 | 44 | 44 | 177
Region of Enrollment [Number; unit: participants]
  France | 12 | 11 | 12 | 12 | 47
  Mexico | 17 | 18 | 18 | 17 | 70
  Belgium | 9 | 7 | 9 | 8 | 33
  Germany | 35 | 37 | 34 | 34 | 140
  Korea, Republic of | 9 | 9 | 9 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Total Severity Score (TSS): Percent Change From Baseline at Week 4
Description: Total Severity Score (TSS) is sum of erythema, scaling and pruritus severity scores of the lesions evaluated each on a 4-point scale from 0 = None to 3 = Severe by the investigator. So minimum TSS can be 0 and maximum 9.
Time Frame: baseline and week 4
Population: Intent To Treat (ITT) with Last Observation Carried Forward (LOCF)
Measure: Median (Full Range); unit: Percent change
Arm/Group | C Propionate 4/Week + Ketoconazole 2/Week | C Propionate 2/Week + Ketoconazole 2/Week | C Propionate 2/Week | Ketakonazol 2/Week
Number analyzed (Participants) | 82 | 82 | 82 | 80
Percent change | -71.4 [-100 to 14.3] | -66.7 [-100 to 0] | -66.7 [-100 to 0] | -57.1 [-100 to 33.3]
Statistical Analysis 1: Comparison: C Propionate 2/Week + Ketoconazole 2/Week vs Ketakonazol 2/Week; The primary efficacy criterion was analyzed by using the Cochran-Mantel-Haenszel (CMH) statistic, stratified by center (or analysis-center) after ridit transformation with the row mean difference statistics, testing the hypothesis of equality. The p-value had to be inferior to 0.05 at week 4, in the ITT/LOCF population. PP analysis was also performed to assess the robustness of the results obtained in the ITT/LOCF population; Test type: Superiority or Other; p < 0.01, Cochran-Mantel-Haenszel; Each test was two-sided, at the 0.050 significance level
Statistical Analysis 2: Comparison: C Propionate 2/Week vs Ketakonazol 2/Week; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.039, Cochran-Mantel-Haenszel; Each test was two-sided, at the 0.050 significance level

ADVERSE EVENTS:
Time Frame: During the study - 12 weeks
Arm/Group | C Propionate 4/Week + Ketoconazole 2/Week | C Propionate 2/Week + Ketoconazole 2/Week | C Propionate 2/Week | Ketakonazol 2/Week
Serious Adverse Events (participants affected / at risk) | 1/82 | 0/82 | 1/82 | 0/80
Other Adverse Events (participants affected / at risk) | 15/82 | 18/82 | 17/82 | 16/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C Propionate 4/Week + Ketoconazole 2/Week (N=82) | C Propionate 2/Week + Ketoconazole 2/Week (N=82) | C Propionate 2/Week (N=82) | Ketakonazol 2/Week (N=80)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C Propionate 4/Week + Ketoconazole 2/Week (N=82) | C Propionate 2/Week + Ketoconazole 2/Week (N=82) | C Propionate 2/Week (N=82) | Ketakonazol 2/Week (N=80)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dymenorrhoea (Reproductive system and breast disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Influenza (Infections and infestations) | 3 (3) | 4 (4) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (6) | 4 (4) | 7 (7) | 5 (7)
Pharyngitis (Infections and infestations) | 2 (3) | 1 (1) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any intent of the investigator to publish or disclose in any way the information requires the sponsor's prior written approval. The investigator shall provide their draft of such publication to sponsor to review and approval at least 2 months prior to the date of intended publication. Sponsor shall have the absolute right to determine whether information may be published by the investigator.